CLINICAL TRIAL: NCT01688869
Title: Mild Traumatic Brain Injury Registry
Acronym: mTBI
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 04-12-03A
Record Dates: First submitted 2012-09-17; First posted 2012-09-20 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2015-02

CONDITIONS: Brain Injury, Traumatic
Keywords: brain concussion
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be obtained in the emergency room and processed for future analysis. Depending on the blood volume obtained, up to two citrate, two EDTA, and one Paxgene tube will be collected.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Mild TBI: Patients who have been diagnosed with a mild brain injury.

SUMMARY:
The purpose of the study is to gather information about patients with mild traumatic brain injury in order to develop guidelines for evaluation and treatment.

DETAILED DESCRIPTION:
The Mild Traumatic Brain Injury Registry is a prospective study which includes patients who have been seen in the CMC ED with a diagnosis of mild brain injury or concussion and a negative CT scan. The investigators will be collecting blood samples, and administering cognitive and balance tests. The investigators will also be following symptoms and cognition throughout the first year to help define typical recovery, and guide prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Must have defined history of CHI (closed head injury) which produced an altered state of consciousness or mood
* Must be awake and alert (Glasgow Coma Scale 13-15)
* Must be enrolled within 72 hours of injury
* Must have CT or MRI neuroimaging performed

Exclusion Criteria:

* Diabetes Mellitus with severe complications
* Intoxication at time of enrollment
* Major psychiatric disorder that is poorly controlled
* Prior stroke
* History of Social Security defined "disability
* Uncontrolled Seizure Disorder
* Incarceration or arrest
* Concurrent Injury requiring hospitalization
* Use of anticoagulant drugs
* Any condition the investigator deems as inappropriate for patient enrollment
* Personality disorder
* Heart, liver or kidney failure defined using common clinical practice guidelines
* Baseline cognitive impairment
* Homelessness
* TBI associated with interpersonal violence
* Pregnancy
* Long bone fracture requiring surgical stabilization

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who are seen in the CMC emergency department who have a clearly defined history of traumatic brain injury that produced at least transient alteration in consciousness, or change in mood, together with one or more persistent symptom lasting longer than one hour after impact. Symptoms can include head pain, nausea, dizziness, disequilibrium, confusion, amnesia, or irritability. All patients must be awake and alert (GCS 13 to 15), and must be enrolled within 72 hours of the injury.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
To determine which biomarkers and/or clinical variables correlate with long term symptoms of mild traumatic brain injury. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lori M Grafton, MD, Principal Investigator — Wake Forest University Health Sciences; Michael A Gibbs, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States